CLINICAL TRIAL: NCT02015676
Title: 'A Study of the Effect of First Line Treatment With Paclitaxel and Myocet in Combination With Herceptin on Overall Tumor Response in Patients With Metastatic or Locally Advanced Breast Cancer and HER2 Overexpression.'
Brief Title: A Study of Herceptin (Trastuzumab) in Combination Chemotherapy in Patients With Metastatic or Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M77035
Record Dates: First submitted 2013-12-03; First posted 2013-12-19 (Estimated); Results first posted 2015-03-12 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Paclitaxel; Doxorubicin

ARMS (2):
- Trastuzumab, Myocet, Paclitaxel; Phase I (Experimental): Participants received an initial loading dose of trastuzumab 4 milligrams per kilogram (mg/kg), intravenously (IV), over 1.5 hours during Week 1, followed by 2 mg/kg, IV, over 30 minutes once per week from Week 2 to Week 52 or until disease progression. Participants also received myocet, 40 mg/ square meter (m^2), IV, every 3 weeks, from Week 1; if no dose limiting toxicity (DLT) was observed in greater than or equal to (≥) two-thirds (2/3) of cohort for 2 treatment cycles, the dose was increased to 50 mg/m^2, IV, and continued for 6 cycles. Participants also received paclitaxel 60 mg/ m^2, IV, once per week, from Week 19; if no DLT was observed in ≥ 2/3 of cohort for 2 treatment cycles, the dose was increased to 70 mg/m^2, IV, and subsequently 80 mg/m^2, IV, and continued until disease progression.
  Interventions: Drug: trastuzumab; Drug: paclitaxel; Drug: Myocet
- Trastuzumab, Myocet, Paclitaxel; Phase II (Experimental): Participants received an initial loading dose of trastuzumab 4 mg/kg, IV, over 1.5 hours during Week 1, followed by 2 mg/kg, IV, over 30 minutes once per week from Week 2 to Week 52 or until disease progression. Participants also received myocet, 50 mg/m^2, IV, every 3 weeks, from Week 1 for 6 cycles. Participants also received paclitaxel 80 mg/m^2, IV, once per week, from Week 19 until disease progression.
  Interventions: Drug: trastuzumab; Drug: paclitaxel; Drug: Myocet

INTERVENTIONS:
Drug: trastuzumab — Initial loading does of 4 mg/kg IV, followed by 2 mg/kg IV weekly, until disease progression
  Other Names: Herceptin
Drug: paclitaxel — 60 mg/m^2 IV weekly; dose increased to 70 mg/m^2, and subsequently 80 mg/m^2, after 2 treatment cycles with no evidence of DLT until disease progression
Drug: Myocet — 40 mg/m^2 IV weekly; dose increased to 50 mg/m^2 IV after 2 treatment cycles with no evidence of DLT for 6 cycles

SUMMARY:
This study will define an optimal chemotherapy dose regimen of Myocet in combination with paclitaxel and intravenous Herceptin and will evaluate the efficacy and safety of this dose regimen in patients with metastatic or locally advanced breast cancer and HER2 overexpression. The anticipated time on study treatment is 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* women 18-70 years of age;
* metastatic or locally advanced breast cancer;
* HER2 overexpression;
* >= 1 measurable lesion.

Exclusion Criteria:

* prior treatment for advanced breast cancer;
* prior treatment with Herceptin;
* bone or central nervous system metastasis as the only site of disease;
* history of another malignancy (except basal cell skin cancer and cancer in situ of the uterine cervix, and contralateral breast cancer) within 5 years of study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2001-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (1):
- Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab, Doxorubicin, Paclitaxel; Phase I: Participants received an initial loading dose of trastuzumab 4 milligrams per kilogram (mg/kg), intravenously (IV), over 1.5 hours on Day 1 (Week 1), followed by 2 mg/kg, IV, over 30 minutes once per week from Week 2 to Week 52 or until disease progression; doxorubicin, 40 mg per square meter (mg/m^2), IV, once every 3 weeks, from Week 1. If no dose-limiting toxicity (DLT) was observed in greater than or equal to (≥) two-thirds (2/3) of cohort for 2 treatment cycles, the dose was increased to 50 mg/m^2, IV, and continued for 6 cycles; and paclitaxel 60 mg/m^2, IV, once per week, starting at Week 19; if no DLT was observed in ≥2/3 of cohort for 2 treatment cycles, the dose was increased to 70 mg/m^2, IV, and subsequently 80 mg/m^2, IV, and continued until disease progression.
- Trastuzumab, Doxorubicin, Paclitaxel; Phase II: Participants received an initial loading dose of trastuzumab 4 mg/kg, IV, over 1.5 hours on Day 1 (Week 1), followed by 2 mg/kg, IV, over 30 minutes once per week from Week 2 to Week 52 or until disease progression; doxorubicin, 50 mg/m^2, IV, once every 3 weeks, starting at Week 1 for 6 cycles; and paclitaxel 80 mg/m^2, IV, once per week, from Week 19 until disease progression.
- Trastuzumab Doxorubicin, Paclitaxel; Phase I and Phase II: During Phase I, participants received an initial loading dose of trastuzumab 4 mg/kg, IV, over 1.5 hours on Day 1 (Week 1), followed by 2 mg/kg, IV, over 30 minutes once per week from Week 2 to Week 52 or until disease progression; doxorubicin, 40 mg/m^2, IV, once every 3 weeks, for 2 treatment cycles, then the dose was increased to 50 mg/m^2, IV, and continued for 6 cycles; and paclitaxel 60 mg/m^2, IV, once per week, starting at Week 19 for 2 treatment cycles, then the dose was increased to 70 mg/m^2, IV, and subsequently 80 mg/m^2, IV, and continued until disease progression. In Phase II, participants received an initial loading dose of trastuzumab 4 mg/kg, IV, over 1.5 hours on Day 1 (Week 1), followed by 2 mg/kg, IV, over 30 minutes once per week from Week 2 to Week 52 or until disease progression; doxorubicin, 50 mg/m^2, IV, once every 3 weeks, starting at Week 1 for 6 cycles; and paclitaxel 80 mg/m^2, IV, once per week, from Week 19 until disease progression.
Period: Overall Study
Arm/Group | Trastuzumab, Doxorubicin, Paclitaxel; Phase I | Trastuzumab, Doxorubicin, Paclitaxel; Phase II | Trastuzumab Doxorubicin, Paclitaxel; Phase I and Phase II
Started | 15 | 48 | 6
Completed | 6 | 14 | 3
Not Completed | 9 | 34 | 3
Not completed — Adverse Event | 2 | 18 | 0
Not completed — Lack of Efficacy | 2 | 4 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 7 | 1
Not completed — Administrative reasons | 0 | 3 | 1
Not completed — Death | 0 | 1 | 0
Not completed — Disease progression | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Trastuzumab, Doxorubicin, Paclitaxel; Phase I: Participants received an initial loading dose of trastuzumab 4 mg/kg, IV, over 1.5 hours on Day 1 (Week 1), followed by 2 mg/kg, IV, over 30 minutes once per week from Week 2 to Week 52 or until disease progression; doxorubicin, 40 mg/m^2, IV, once every 3 weeks, from Week 1. If no DLT was observed in ≥2/3 of cohort for 2 treatment cycles, the dose was increased to 50 mg/m^2, IV, and continued for 6 cycles; and paclitaxel 60 mg/m^2, IV, once per week, starting at Week 19; if no DLT was observed in ≥2/3 of cohort for 2 treatment cycles, the dose was increased to 70 mg/m^2, IV, and subsequently 80 mg/m^2, IV, and continued until disease progression.
- Trastuzumab, Doxorubicin, Paclitaxel; Phase II and II: During Phase I, participants received an initial loading dose of trastuzumab 4 mg/kg, IV, over 1.5 hours on Day 1 (Week 1), followed by 2 mg/kg, IV, over 30 minutes once per week from Week 2 to Week 52 or until disease progression; doxorubicin, 40 mg/m^2, IV, once every 3 weeks, for 2 treatment cycles, then the dose was increased to 50 mg/m^2, IV, and continued for 6 cycles; and paclitaxel 60 mg/m^2, IV, once per week, starting at Week 19 for 2 treatment cycles, then the dose was increased to 70 mg/m^2, IV, and subsequently 80 mg/m^2, IV, and continued until disease progression. In Phase II, participants received an initial loading dose of trastuzumab 4 mg/kg, IV, over 1.5 hours on Day 1 (Week 1), followed by 2 mg/kg, IV, over 30 minutes once per week from Week 2 to Week 52 or until disease progression; doxorubicin, 50 mg/m^2, IV, once every 3 weeks, starting at Week 1 for 6 cycles; and paclitaxel 80 mg/m^2, IV, once per week, from Week 19 until disease progression.
- Total: Total of all reporting groups
Arm/Group | Trastuzumab, Doxorubicin, Paclitaxel; Phase I | Trastuzumab, Doxorubicin, Paclitaxel; Phase II | Trastuzumab, Doxorubicin, Paclitaxel; Phase II and II | Total
Number analyzed (Participants) | 15 | 48 | 6 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.73 (12.42) | 52.98 (12.33) | 44.33 (15.36) | 52.61 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 48 | 6 | 69
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) According to World Health Organization (WHO) Handbook for Reporting Results of Cancer Treatment
Description: For measurable disease, CR was defined as the disappearance of all clinically detectable disease determined by 2 observations not less than 4 weeks apart; and PR was defined as a 50 percent (%) decrease in the sum of the products of the 2 greatest diameters of all measurable lesions by 2 observations not less than 4 weeks apart, and no appearance of new lesions or progression of any lesion. For immeasurable disease, CR was defined as the complete disappearance of all known disease for at least 4 weeks; and PR was defined as an estimated decrease in tumor size of 50% or more for at least 4 weeks.
Time Frame: Baseline (BL), Weeks 7, 13, 19, every 8 weeks thereafter until end of study (for up to 3 years)
Population: All participants enrolled in Phase II of this study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab, Doxorubicin, Paclitaxel; Phase II
Number analyzed (Participants) | 54
percentage of participants
  CR | 51.85
  PR | 46.30

2. Secondary Outcome: Time to Disease Progression - Percentage of Participants With an Event
Description: Disease progression was defined as the time from the start of treatment to the date of the first recorded incident of disease progression, or the date of death due any cause. For measurable disease, disease progression was defined as a ≥25% increase in the sum of the products of diameters of 1 or more measurable lesions with a minimal area of greater than (>)2 square centimeters (cm^2), or the appearance of new lesions; and for malignant lesions with a minimal area of 2 cm^2, an increase of ≥1 cm^2. For immeasurable disease, disease progression was defined as the appearance of any new lesion not previously identified or an estimated increase of ≥50% in existent lesions.
Time Frame: BL, Weeks 7, 13, 19, every 8 weeks thereafter until end of study (for up to 3 years)
Population: All participants enrolled in Phase II of this study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab, Doxorubicin, Paclitaxel; Phase II
Number analyzed (Participants) | 54
percentage of participants | 40.74

3. Secondary Outcome: Time to Disease Progression
Description: The median time, in months, from the start of treatment to disease progression event.
Time Frame: BL, Weeks 7, 13, 19, every 8 weeks thereafter until end of study (for up to 3 years)
Population: All participants enrolled in Phase II of this study were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab, Doxorubicin, Paclitaxel; Phase II
Number analyzed (Participants) | 54
months | 43.3018 [24.0821 to NA] — Upper limit of the 95% confidence interval (CI) could not be estimated because the largest observation was censored and the estimation was restricted to the largest event time.

4. Secondary Outcome: Time to Treatment Response - Percentage of Participants With an Event
Description: Treatment response was defined as the time from the start of treatment to the date of recorded CR or PR of measurable disease.
Time Frame: BL, Weeks 7, 13, 19, every 8 weeks thereafter until end of study (for up to 3 years)
Population: All participants enrolled in Phase II of this study were included in the analysis.
Measure: Number; unit: percentage participants
Arm/Group | Trastuzumab, Doxorubicin, Paclitaxel; Phase II
Number analyzed (Participants) | 54
percentage participants | 98.15

5. Secondary Outcome: Time to Treatment Response
Description: The median time, in months, from the start of treatment to treatment response event.
Time Frame: BL, Weeks 7, 13, 19, every 8 weeks thereafter until end of study (for up to 3 years)
Population: All participants enrolled in Phase II of this study were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab, Doxorubicin, Paclitaxel; Phase II
Number analyzed (Participants) | 54
months | 1.87269 [1.83984 to 1.93840]

6. Secondary Outcome: Duration of Response - Percentage of Participants With an Event
Description: Duration of response was defined as the time from date CR was first recorded to the date progressive disease (PD) was first noted. For measurable disease, PD was defined as a ≥25% increase in the sum of the products of diameters of 1 or more measurable lesions with a minimal area of >2 cm^2, or the appearance of new lesions; and for malignant lesions with a minimal area of 2 cm^2, an increase of ≥1 cm^2. For immeasurable disease, PD was defined as the appearance of any new lesion not previously identified or an estimated increase of ≥50% in existent lesions.
Time Frame: BL, Weeks 7, 13, 19, every 8 weeks thereafter until end of study (for up to 3 years)
Population: Only participants with a response were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab, Doxorubicin, Paclitaxel; Phase II
Number analyzed (Participants) | 53
percentage of participants | 39.62

7. Secondary Outcome: Duration of Response
Description: The median time, in months, from enrollment to duration of response event to Week 52.
Time Frame: BL, Weeks 7, 13, 19, every 8 weeks thereafter until end of study (for up to 3 years)
Population: All participants enrolled in Phase II of this study were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab, Doxorubicin, Paclitaxel; Phase II
Number analyzed (Participants) | 54
months | 41.1006 [20.9610 to NA] — Upper limit of the 95% CI could not be estimated because the largest observation was censored and the estimation was restricted to the largest event time.

8. Secondary Outcome: Time to Therapy Failure - Percentage of Participants With an Event
Description: Therapy failure was defined as the date of the start of therapy to the date of withdrawal due to adverse events, progressive disease/insufficient therapeutic response, death, failure to return, or refusal of treatment/lack of cooperation/withdrawal of consent. Participants were censored at the last dose of treatment if no event was recorded.
Time Frame: BL, Weeks 7, 13, 19, every 8 weeks thereafter until end of study (for up to 3 years)
Population: All participants enrolled in Phase II of this study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab, Doxorubicin, Paclitaxel; Phase II
Number analyzed (Participants) | 54
percentage of participants | 81.48

9. Secondary Outcome: Time to Therapy Failure
Description: The median time, in months, from treatment start to therapy failure event. Participants were censored at the last date of treatment if no event was recorded.
Time Frame: BL, Weeks 7, 13, 19, every 8 weeks thereafter until end of study (for up to 3 years)
Population: All participants enrolled in Phase II of this study were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab, Doxorubicin, Paclitaxel; Phase II
Number analyzed (Participants) | 54
months | 24.0821 [17.5113 to 35.6797]

10. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With an Event
Description: OS was defined as the time from the date of the start of treatment to the date of death or the last date the participant was known to be alive.
Time Frame: BL, Weeks 7, 13, 19, every 8 weeks thereafter until end of study (for up to 3 years)
Population: All participants enrolled in Phase II of this study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab, Doxorubicin, Paclitaxel; Phase II
Number analyzed (Participants) | 54
percentage of participants | 3.70

11. Secondary Outcome: Overall Survival
Description: The time, in months, from the start of treatment to OS event. The mean survival time and it's standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time.
Time Frame: BL, Weeks 7, 13, 19, every 8 weeks thereafter until end of study (for up to 3 years)
Population: All participants enrolled in Phase II of this study were included in the analysis.
Measure: Mean (Standard Error); unit: months
Arm/Group | Trastuzumab, Doxorubicin, Paclitaxel; Phase II
Number analyzed (Participants) | 54
months | 7.6909 (0.1338)

ADVERSE EVENTS:
Time Frame: BL, and Weeks 7, 13, 19, every 8 weeks thereafter until end of study.
Description: All participants who received at least 1 dose of study treatment and at least 1 safety follow-up were included in the safety analysis.
Groups:
- Trastuzumab, Doxorubicin, Paclitaxel; Phase I & II: Participants received an initial loading dose of trastuzumab 4 mg/kg, IV, over 1.5 hours on Day 1 (Week 1), followed by 2 mg/kg, IV, over 30 minutes once per week from Week 2 to Week 52 or until disease progression; doxorubicin, 50 mg/m^2, IV, once every 3 weeks, starting at Week 1 for 6 cycles; and paclitaxel 80 mg/m^2, IV, once per week, from Week 19 until disease progression.
Arm/Group | Trastuzumab, Doxorubicin, Paclitaxel; Phase I & II
Serious Adverse Events (participants affected / at risk) | 26/69
Other Adverse Events (participants affected / at risk) | 63/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab, Doxorubicin, Paclitaxel; Phase I & II (N=69)
Febrile neutropenia (General disorders) | 12
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intestinal obstruction NOS (Gastrointestinal disorders) | 1
Cardiac failure NOS (Cardiac disorders) | 2
Endocarditis (Infections and infestations) | 1
Pancreatitis NOS (Infections and infestations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Diarrhoea NOS (Gastrointestinal disorders) | 2
Skin infection (Skin and subcutaneous tissue disorders) | 1
Pancreatitis (Infections and infestations) | 1
Respiratory tract infection NOS (Infections and infestations) | 1
Pneumonia NOS (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory tract infection NOS (Infections and infestations) | 1
Thrombophlebitis (Blood and lymphatic system disorders) | 1
Anaemia NOS (Blood and lymphatic system disorders) | 1
Acute febrile neutrophilic dermatosis (Blood and lymphatic system disorders) | 1
Staphylococcal infection (Infections and infestations) | 1
Ejection fraction decreased (Cardiac disorders) | 1
Mucosal inflammation NOS (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab, Doxorubicin, Paclitaxel; Phase I & II (N=69)
Abdominal pain NOS (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 11
Alopecia (Skin and subcutaneous tissue disorders) | 54
Amenorrhoea NOS (Reproductive system and breast disorders) | 9
Anaemia NOS (Blood and lymphatic system disorders) | 7
Anal fissure (Gastrointestinal disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 10
Anxiety symptoms (Psychiatric disorders) | 2
Aphonia (Nervous system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Asthenia (General disorders) | 35
Back pain (Musculoskeletal and connective tissue disorders) | 15
Biliary colic (Hepatobiliary disorders) | 1
Blood bilirubin increased (Investigations) | 1
Body tinea (Skin and subcutaneous tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 6
Bowel sounds abnormal (Gastrointestinal disorders) | 1
Breast abscess (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast pain (Reproductive system and breast disorders) | 2
Bronchitis NOS (Respiratory, thoracic and mediastinal disorders) | 2
Bronchospasm NOS (Respiratory, thoracic and mediastinal disorders) | 1
Cardiotoxicty (Cardiac disorders) | 2
Catarrh (General disorders) | 5
Catheter related infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cheilitis (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 3
Chest wall pain (General disorders) | 2
Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Conjunctivitis (Eye disorders) | 11
Constipation (Gastrointestinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Cystitis-like symptom (Renal and urinary disorders) | 1
Death NOS (General disorders) | 1
Depression (Psychiatric disorders) | 8
Dermatitis NOS (Skin and subcutaneous tissue disorders) | 1
Dermatitis radiation NOS (Skin and subcutaneous tissue disorders) | 7
Diarrhoea NOS (Gastrointestinal disorders) | 29
Dizziness (Nervous system disorders) | 5
Drug hypersensitivity (Immune system disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysaesthesia (Nervous system disorders) | 3
Dysgeusia (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 12
Dysphagia (Gastrointestinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Dysuria (Renal and urinary disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Ejection fraction decreased (Cardiac disorders) | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13
Erythema (Skin and subcutaneous tissue disorders) | 13
Extrapyramidal disorder (Nervous system disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 17
Febrile neutropenia (Infections and infestations) | 2
Flushing (Vascular disorders) | 4
Folliculitis (Skin and subcutaneous tissue disorders) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis NOS (Gastrointestinal disorders) | 2
Gingival pain (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemoglobin abnormal (Investigations) | 6
Haemorrhoids (Gastrointestinal disorders) | 6
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 9
Herpes simplex (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hordeolum (Infections and infestations) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypersensitivity NOS (Immune system disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypophonesis (General disorders) | 1
Hypotension NOS (Vascular disorders) | 1
Influenza like illness (General disorders) | 4
Influenza viral infections (Infections and infestations) | 1
Injury asphyxiation (Respiratory, thoracic and mediastinal disorders) | 1
Insomnia (Psychiatric disorders) | 7
Intermittent pyrexia (General disorders) | 1
Intertrigo candida (Metabolism and nutrition disorders) | 1
Joint sprain (Injury, poisoning and procedural complications) | 1
Lacrimation increased (Eye disorders) | 2
Laryngitis NOS (Infections and infestations) | 1
Leukopenia NOS (Blood and lymphatic system disorders) | 3
Limb discomfort NOS (Musculoskeletal and connective tissue disorders) | 1
Lymphangitis (Infections and infestations) | 2
Lymphoedema NOS (Vascular disorders) | 9
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Milk allergy (Immune system disorders) | 1
Mucosal inflammation NOS (Respiratory, thoracic and mediastinal disorders) | 40
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mydriasis (Eye disorders) | 1
Nail discolouration (General disorders) | 1
Nail discomfort (General disorders) | 1
Nail disorder NOS (General disorders) | 23
Nail infection (Infections and infestations) | 1
Nail toxicity (General disorders) | 5
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2
Nasopharyngitis (Infections and infestations) | 3
Nausea (Gastrointestinal disorders) | 36
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Nervousness (Psychiatric disorders) | 1
Neuropathic pain (Nervous system disorders) | 1
Neuropathy NOS (Nervous system disorders) | 5
Neurotoxicity NOS (Nervous system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 21
Not coded (General disorders) | 1
Odynophagia (General disorders) | 3
Oedema NOS (General disorders) | 4
Oedema peripheral (General disorders) | 19
Oesophagitis NOS (Gastrointestinal disorders) | 2
Onycholysis (Skin and subcutaneous tissue disorders) | 9
Oral infection (Infections and infestations) | 2
Oropharyngeal candidiasis (Respiratory, thoracic and mediastinal disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Otitis media NOS (Infections and infestations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pain NOS (General disorders) | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10
Palpitations (Cardiac disorders) | 1
Paraesthesia (Nervous system disorders) | 18
Paralysis (Nervous system disorders) | 1
Paratracheal lymphadenopathy (Blood and lymphatic system disorders) | 1
Performance status decreased (General disorders) | 1
Peripheral neuropathy NOS (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 6
Pharyngitis (Infections and infestations) | 3
Phlebitis NOS (Vascular disorders) | 2
Pigmentation disorder NOS (Skin and subcutaneous tissue disorders) | 4
Pollakiuria (Renal and urinary disorders) | 1
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 1
Post procedural vomiting (Injury, poisoning and procedural complications) | 1
Proctalgia (Gastrointestinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pupils unequal (Eye disorders) | 1
Pyrexia (General disorders) | 23
Rash NOS (Skin and subcutaneous tissue disorders) | 10
Rectal tenesmus (Gastrointestinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Rigors (General disorders) | 7
Scar pain (General disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Sinusitis NOS (Infections and infestations) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 8
Skin infection (Infections and infestations) | 1
Skin reaction (Immune system disorders) | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 5
Stomatitis (Gastrointestinal disorders) | 10
Sweating increased (General disorders) | 1
Syncope (Nervous system disorders) | 2
Tachycardia NOS (Cardiac disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tinea pedis (Infections and infestations) | 1
Toothache (Gastrointestinal disorders) | 1
Transaminases increased (Investigations) | 1
Transient ischaemic attack (Cardiac disorders) | 1
Upper respiratory tract infection NOS (Infections and infestations) | 4
Urinary tract infection NOS (Infections and infestations) | 4
Varicella (Infections and infestations) | 1
Varicophlebitis (Vascular disorders) | 1
Varicose veins NOS (Vascular disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Vision blurred (Eye disorders) | 1
Vomiting NOS (Gastrointestinal disorders) | 26
Weight increased (Investigations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.